CLINICAL TRIAL: NCT06259604
Title: The Effect of Oral Motor Intervention (PIOMI) and Combined Kangaroo Care Applied to Preterm Babies on Weight Gain, Oral Feeding Skills, Transition to Full Oral Feeding and Discharge Time: Randomized Controlled Study
Brief Title: Preterm Infant Oral Motor Intervention (PIOMI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Serife Tutar, Assistant professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 009962
Record Dates: First submitted 2024-01-04; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Feeding Behavior
Keywords: Preterm newborn; Oral feeding; Kangaroo mother care; oral stimulation
MeSH Terms: conditions — Premature Birth; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator
Masking Description: One-sided blinding method will be applied in the research. Only one of the researchers has a PIOMI practitioner certificate and interventions will be carried out only by this researcher. The PIOMI practitioner researcher will perform all interventions of PIOMI and combined methods himself and will not tell other researchers which group the babies are in. All measurements of the babies, except PIOMI, will be carried out by a single researcher in the research group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PIOMI (Experimental): Babies in this group will be administered PIOMI once a day, 30-45 minutes before feeding, for 14 days. When the intervention ends, the baby's feeding will be carried out by the researcher neonatal nurse in a semi-elevated side position, taking into account cue-based feeding symptoms, and the transition to full oral feeding will be evaluated by two researchers. These babies will be evaluated with the Early Feeding Skills Assessment Tool for early feeding skills before any intervention is applied (day 0) and on the 14th day of the PIOMI intervention. In addition, the weight of the babies will be monitored every morning for 14 days, on an empty stomach and naked, and will be recorded in the Nutrition Tracking Chart. The time it takes for babies to transition to full oral feeding will be evaluated according to cue-based feeding and recorded in the Feeding Follow-Up Chart.
  Interventions: Other: PIOMI
- PIOMI+kangaroo care (Experimental): Babies in this group will start using PIOMI once a day, 30-45 minutes before feeding, and kangaroo care for at least 30 minutes during the last 2 minutes of non-nutritive sucking phase of PIOMI, for 14 days. When the intervention ends, the baby's feeding will be carried out by the researcher neonatal nurse in a semi-elevated side position, taking into account cue-based feeding symptoms, and the transition to full oral feeding will be evaluated by two researchers. These babies will be evaluated with the Early Feeding Skills Assessment Tool before any intervention is applied (day 0) and on the 14th day of PIOMI+kangaroo care in terms of early feeding skills. In addition, the weight of the babies will be monitored every morning for 14 days, on an empty stomach and naked, and will be recorded in the Nutrition Tracking Chart. The time it takes for babies to transition to full oral feeding will be evaluated according to cue-based feeding and recorded in the Feeding Follow-Up Chart.
  Interventions: Other: PIOMI+kangaroo care
- Control (No Intervention): Babies in this group will receive standard care in the clinic. They will be evaluated with the Early Nutrition Skills Assessment Tool in terms of early feeding skills on the day they are included in the study (day 0) and on the 14th day. In addition, the weight of the babies will be monitored every morning for 14 days, on an empty stomach and naked, and will be recorded in the Nutrition Tracking Chart. The time it takes for babies to transition to full oral feeding will be evaluated according to cue-based feeding and recorded in the Feeding Follow-Up Chart. All measurements will be carried out and evaluated separately by two independent researchers. During discharge, discharge time, discharge weight and postmenstrual week at discharge will be recorded in the Baby Information Form.

INTERVENTIONS:
Other: PIOMI — Babies in this group will be administered PIOMI once a day, 30-45 minutes before feeding, for 14 days.
  Arms: PIOMI
Other: PIOMI+kangaroo care — Babies in this group will start using PIOMI once a day, 30-45 minutes before feeding, and kangaroo care for at least 30 minutes during the last 2 minutes of non-nutritive sucking phase of PIOMI, for 14 days.
  Arms: PIOMI+kangaroo care

SUMMARY:
The purpose of this research; The aim of this study is to examine the effects of oral motor intervention (PIOMI) and combined kangaroo care applied to preterm babies on weight gain, oral feeding skills, transition to full oral feeding and discharge time.

DETAILED DESCRIPTION:
The most important responsibility for the transition to oral feeding in the early period falls on neonatal intensive care nurses. Neonatal intensive care nurses should evaluate premature babies' readiness for feeding and use evidence-based practices in this regard. Studies show that there are different applications (piomi, fucile, etc.) in oral motor stimulation that provides a single sensory input. One of the most commonly used applications is the PIOMI (Preterm Infant Oral Motor Intervention) application developed by Lessen et al. (2011). PIOMI has been shown to shorten the duration of transition to oral feeding and hospital stay, helps in weight gain, increases sucking capacity and transition from breast to breastfeeding. It is stated that it accelerates the duration. However, PIOMI; such as massage therapy, breastfeeding, oral support and non-nutritive sucking, music therapy. A limited number of studies show that combined use is more effective, and more research is needed in this area.

One of the methods that accelerates the transition to oral feeding in preterm babies and is effective in physiological stability and neuromotor development is kangaroo mother care. No research has been found in the literature examining the effect of kangaroo care and PIOMI application on the oral feeding process of preterm babies when applied in combination. Additionally, no study has been found that evaluated the maturity of oral feeding skills and early feeding skills in which PIOMI and kangaroo care were combined. In this context, research; It will be carried out to examine the effects of oral motor intervention (PIOMI) and combined kangaroo care applied to preterm babies on weight gain, oral feeding skills, transition to full oral feeding and discharge time.

The research is a randomized controlled trial. The research will be carried out in the Neonatal Intensive Care Unit of Isparta City Hospital between March 2024 and March 2025. Neonatal Intensive Care Unit consists of Level 3 with 12 beds, Level 2 with 8 beds, mother-baby adaptation room with 10 beds, 3 isolation rooms and 1 breastfeeding room. There is a breastfeeding nurse at the clinic during the day (8-16) and provides breastfeeding education to mothers. At other times (16-08), each nurse provides breastfeeding counseling to the parents of the baby for whom she/he is responsible for care. Mothers express their milk in the breastfeeding room and hand it over to the nurses, writing the name, date and time on it. Receiving the milked milk to the clinic, storing it and preparing it by heating it. It is carried out in accordance with the Ministry of Health and Food and Drug Administration (FDA). This milk is monitored by each patient's own nurse, and excess milk is put in the freezer. The milk to be used is placed in the milk cabinets in the rooms, and the milk is withdrawn day and night by the nurses according to the doctor's request, before feeding, in accordance with the time, and is heated using the bain-marie method and given to the babies. There is no written protocol in the clinic regarding the transition and maintenance of oral feeding of newborns. Oral feeding is initiated by the joint decision of the neonatal physician and neonatal nurse, taking into account the postmenstrual week, physiological parameters and individual conditions of the newborns. In oral feeding of preterm babies, syringes are generally used and babies are fed in a semi-elevated position.

The data of the research will be collected with the "Informed Volunteer Consent Form", "Baby Introduction Form", "Early Feeding Skills Assessment Tool" and "Nutrition Tracking Chart".

There are three groups in the research: PIOMI, PIOMI+kangaroo care and control group.

One-sided blinding method will be applied in the research. Only one of the researchers has a PIOMI practitioner certificate and interventions will be carried out only by this researcher. The PIOMI practitioner researcher will perform all interventions of PIOMI and combined methods himself and will not tell other researchers which group the babies are in. All measurements of the babies, except PIOMI, will be carried out by a single researcher in the research group.

The data obtained in the research will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods (number, percentage, min-max values, mean, standard deviation) will be used when evaluating the data. Cronbach Alpha values will be calculated to test the reliability of the scales used in the research. The compliance of continuous variables used in the research with normal distribution will be determined. Compliance with normal distribution can be examined in 3 different ways. Compliance with normal distribution can be determined by analyzing it with Shapiro Wilk or Kolmogrov Simrnov tests. It can also be examined by drawing a Q-Q plot. In this method, the normal distribution of the data used will be checked by checking whether the skewness and kurtosis values are between ±3.

Parametric tests will be used in statistical evaluations for variables with normal distribution. In comparing quantitative data on variables with normal distribution, independent t test determines the difference between two groups; F test for more than two groups; Non-parametric tests will be used in statistical evaluations for variables that do not have a normal distribution. In comparing quantitative data on scales that do not have a normal distribution, the Mann Whitney U test determines the difference between two groups; For more than two groups, the Kruskal Wallis H test will be applied. Dependent sample tests will be used to examine the changes within groups. Dependent sample t test on normally distributed data; For data that does not show normal distribution, the Wilcoxon sign test will be used. Intraclass correlation coefficient (ICC) will be calculated to evaluate interobserver agreement.

In order to conduct this research, approval will be obtained from the Süleyman Demirel University Faculty of Medicine Clinical Research Ethics Committee. In addition, institutional permission will be obtained from the hospital where the research is planned to be conducted and written informed consent will be obtained from the parents of the babies included in the research. Permission for the PIOMI application was obtained via e-mail from Brenda Lessen Knoll.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth is 28-32 weeks, depending on the mother's last menstrual period,
* 29-32. can be administered PIOMI per week and can tolerate the transition to oral feeding,
* Able to tolerate the transition to oral feeding according to the cue-based feeding model,
* Maintains physiological stabilization (heart rate, oxygen saturation, respiratory rate) during the procedure when oxygen support is provided with room air or nasal cannula or hood.
* Apgar score of 4 or higher at the 5th minute after birth
* Not receiving mechanical ventilator support or 48 hours after weaning from mechanical ventilator support
* Babies with written and verbal permission from their parents will be included in the research.

Exclusion Criteria:

* Those with congenital anomalies (cleft lip, cleft palate, gastroschisis, omphalocele, short bowel syndrome and other anomalies) According to the criteria of Jobe and Bancalari (2001), patients with severe bronchopulmonary dysplasia and patent ductus arteriosus (PDA) requiring surgical treatment Babies with gastrointestinal, neurological and genetic diseases (necrotizing enterocolitis, level 3 and 4 intracranial hemorrhage, periventricular 25 leukomalacia, hydrocephalus, down syndrome) will not be included in the study.

Ages: 29 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
weight change | Up to 14 days
  The baby's weight chage will be recorded.
Early Feeding Skills Assessment Tool Scores | Before the intervention and on the 14th day of the intervention. The overall Early Feeding Skills Assessment Tool score is the sum of the 5 subscale scores and ranges from 19 to 57. Higher scores indicate more mature feeding skills.
  Oral motor control will be evaluated.
Transition time to full oral feeding | Up to 14 days
  The baby's transition to full oral feeding will be recorded.
Discharge period | through the baby's hospital admission to discharge
  The time from hospital admission to discharge will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Tutar, Dr., Principal Investigator — Suleyman Demirel University
Locations (1):
- Isparta City Hospital, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After our research is completed, the research results will be shared with other researchers.